CLINICAL TRIAL: NCT01032564
Title: Interest of HI-RTE Elasticity in Obstetric
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2009-A00814-53; 2009-22
Record Dates: First submitted 2009-12-11; First posted 2009-12-15 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Premature Birth
Keywords: estimate the interest of the measure of cervix elasticity degree by elastography in prediction of premature birth within a population of pregnant women
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: The elastography (elasticity imagery) — This diagnosis mean use the ultrasonography to measure the tissues answer under pressure

SUMMARY:
In obstetric, the investigators can't predict accurately with current means (BISHOP score, traditional cervix ultrasonography and fibronectin) the childbirth time and delay.

If ultrasonography can determine the length, the cervix opening, it can't define its flexibility. Indeed, the conventional cervix ultrasonography can't inform us about the consistency of the uterine cervix.

The elastography (elasticity imagery) is an innovating technology. It is a new technology currently used as part of breast cancer estimate. This diagnosis mean use the ultrasonography to measure the tissues answer under pressure.

Its contribution in obstetric must be estimated to improve patients minimum fare.

The main target of the investigators study is to estimate the interest of the measure of cervix elasticity degree by elastography in prediction of premature birth within a population of pregnant women

ELIGIBILITY:
Inclusion Criteria:

* Unique(only) or multiple pregnancy about is the term presenting an intra Utérine pregnancy in the 1st quarter ·
* Signed lit(enlightened) consent ·
* Patient of more than 18 years old

Exclusion Criteria:

* Suspicion of pregnancy extra utérine, hémodynamique unstable, important métrorragies, maternal diabetes, arterial high blood pressure

  * impossibility to receive the consent lit(enlightened) by the patient · patient old under age 18

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2009-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
The elastography (elasticity imagery) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Florence BRETELLE, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Sabiani L, Haumonte JB, Loundou A, Caro AS, Brunet J, Cocallemen JF, D'ercole C, Bretelle F. Cervical HI-RTE elastography and pregnancy outcome: a prospective study. Eur J Obstet Gynecol Reprod Biol. 2015 Mar;186:80-4. doi: 10.1016/j.ejogrb.2015.01.016. Epub 2015 Jan 23. PMID 25666343